CLINICAL TRIAL: NCT00552071
Title: Study to Determine Whether Ultrasound Guidance Improves Delivery and Efficacy of Intramuscular Injection of Long-Acting Octreotide in the Treatment of Acromegaly
Brief Title: Ultrasound Guided Octreotide LAR Injection in Acromegaly
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cedars-Sinai Medical Center (Other)
Collaborators: Novartis Pharmaceuticals (Industry)
Responsible Party: Principal Investigator, John Carmichael, Co Director, Pituitary Program At Keck Medical Center, University of Southern California
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 11482; CSMS995BUS60 (Other: Other)
Record Dates: First submitted 2007-10-31; First posted 2007-11-01 (Estimated); Results first posted 2018-09-11 (Actual); Last update posted 2018-09-11 (Actual); Status verified 2018-08

CONDITIONS: Acromegaly
Keywords: Acromegaly; Octreotide LAR; Ultrasound guidance
MeSH Terms: conditions — Acromegaly | interventions — Injections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Ultrasound-guided IM injections of octreotide LAR (Experimental): Subjects received octreotide LAR 30 mg injection via ultrasound-guided IM gluteal injection every 28 days for 3 months.
  Interventions: Drug: Octreotide LAR 30 MG Injection
- Regular IM injections of octreotide LAR (Active Comparator): Subjects received octreotide LAR 30 mg injection via regular IM gluteal injections every 28 days for 3 months
  Interventions: Drug: Octreotide LAR 30 MG Injection

INTERVENTIONS:
Drug: Octreotide LAR 30 MG Injection — Stable dose of 30 mg octreotide LAR, or a dose determined by historical dosing, delivered every 28 days for 3 months.
  Other Names: Sandostatin LAR

SUMMARY:
Approximately half of patients with acromegaly do not respond to treatment with somatostatin receptor ligands such as octreotide LAR. This may be due to inadequate drug delivery if the standard of care regular injection is inaccurately delivered in the intramuscular (IM) compartment. Ultrasound guidance of IM injections may improve accuracy of placement of IM injections and increase drug levels, thereby improving efficacy of octreotide LAR for the treatment of acromegaly. The purpose of this study is to determine whether octreotide LAR drug levels differ if given by ultrasound-guided IM injection or by regular IM injection in patients with acromegaly.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of active acromegaly based on evidence of a pituitary tumor
* Historical serum insulin-like growth factor (IGF)-I levels or a lack of suppression of growth hormone (GH) < 1 ng/mL during an oral glucose tolerance test
* Previous treatment with a stable dose of octreotide LAR for at least 3 months
* No previous treatment with a stable dose of octreotide LAR for at least 3 months after receiving 3 months of octreotide LAR during a run-in phase prior to any other study-related activity

Exclusion Criteria:

* Uncontrolled diabetes mellitus
* Pregnant or breast feeding
* Current gallstones
* History of hepatic disease, except patients with < 3 X ULN LFTs indicative of hepatic steatosis
* Past or current history of cancer, except for basal cell carcinoma or in situ cancer of the cervix
* History of glucocorticoid therapy within the past 6 months, current treatment with any chemotherapeutic agents or exogenous GH therapy
* History of investigational drugs administered or received within 30 days of study entry
* Known hypersensitivity to octreotide LAR
* Any other concomitant illnesses or therapy that would interfere with evaluation of efficacy or safety or increase the risk for study interruption or discontinuation in the opinion of the investigator or sponsor

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2007-07; Primary Completion 2014-03 (Actual); Study Completion 2014-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: John Carmichael, MD, Principal Investigator — University of Southern California
Locations (1):
- Cedars-Sinai Medical Center, Los Angeles, California, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This study recruited subjects with active acromegaly. Equal numbers of men and women were to be recruited, but the recruitment plan was adjusted during the course of the trial to account for the high number of women withdrawn from the study. 12 women and 9 men were recruited; 8 men and 7 women completed the study and were included in the analysis.
Pre-assignment Details: Subjects who had not received 3 monthly injections of a stable dose of octreotide LAR prior to enrollment were given 3 monthly injections of octreotide LAR at a stable dose of 30 mg every 28 days or at a dose determined by historical dosing. Nine of the 15 subjects participated in this run-in period.
Groups:
- Ultrasound-guided Injections Followed by Regular Injections: Subjects received octreotide LAR via ultrasound-guided IM gluteal injections every 28 days for 3 months followed by regular IM gluteal injections every 28 days for 3 months.
- Regular Injections Followed by Ultrasound-guided Injections: Subjects received octreotide LAR via regular IM gluteal injections every 28 days for 3 months followed by ultrasound-guided IM gluteal injections every 28 days for 3 months.
Period: Overall Study
Arm/Group | Ultrasound-guided Injections Followed by Regular Injections | Regular Injections Followed by Ultrasound-guided Injections
Started | 10 | 11
Completed | 6 | 9
Not Completed | 4 | 2
Not completed — Adverse Event | 1 | 0
Not completed — Lack of Efficacy | 1 | 0
Not completed — Physician Decision | 1 | 0
Not completed — Pregnancy | 1 | 0
Not completed — Death | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ultrasound-guided Injections Followed by Regular Injections | Regular Injections Followed by Ultrasound-guided Injections | Total
Number analyzed (Participants) | 6 | 9 | 15
Age, Continuous [Mean (Standard Deviation); unit: years] | 56 (14) | 53 (16) | 53 (15)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 5 | 7
  Male | 4 | 4 | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 6 | 9 | 15

OUTCOME MEASURES:

1. Primary Outcome: Plasma Octreotide Level After Each Treatment Phase
Description: Venous sampling was performed at each visit immediately prior to each IM injection. Levels were measured at each visit and mean for the group was calculated after each treatment phase.
Time Frame: 3 months
Population: Subjects were regrouped for analysis by treatment. Octreotide levels after 3 monthly octreotide LAR injections with ultrasound guidance were compared to octreotide levels obtained after 3 monthly octreotide LAR injection without ultrasound guidance.
Measure: Mean (Standard Deviation); unit: pg/mL
Groups:
- Ultrasound-guided Injections of Octreotide LAR: All subjects receiving ultrasound-guided injections during the study.
- Regular Injections of Octreotide LAR: All subjects receiving regular injections during the study.
Arm/Group | Ultrasound-guided Injections of Octreotide LAR | Regular Injections of Octreotide LAR
Number analyzed (Participants) | 15 | 15
pg/mL | 885 (702) | 1167 (1126)
Statistical Analysis 1: Comparison: Ultrasound-guided Injections of Octreotide LAR vs Regular Injections of Octreotide LAR; Test type: Other; p = 0.40, t-test, 2 sided — A two-sided p value of <0.05 was considered significant

2. Secondary Outcome: Serum IGF-1 Level
Description: as for outcome 1
Time Frame: 3 months
Population: Subjects were regrouped for analysis by treatment. Serum IGF-I levels after 3 monthly octreotide LAR injections with ultrasound guidance were compared to Serum IGF-I levels obtained after 3 monthly octreotide LAR injection without ultrasound guidance.
Measure: Mean (Standard Deviation); unit: percentage of upper limit of normal
Groups:
- Ultrasound-guided Injections of Octreotide LAR: All subjects who recieved ultrasound-guided injections during the study.
- Regular Injections of Octreotide LAR: All subjects who received regular injections during the study.
Arm/Group | Ultrasound-guided Injections of Octreotide LAR | Regular Injections of Octreotide LAR
Number analyzed (Participants) | 15 | 15
percentage of upper limit of normal | 132 (92) | 124 (83)
Statistical Analysis 1: Comparison: Ultrasound-guided Injections of Octreotide LAR vs Regular Injections of Octreotide LAR; Test type: Other; p = 0.43, t-test, 2 sided — A two-sided p value of <0.05 was considered significant

ADVERSE EVENTS:
Time Frame: 6 months
Description: Arms/Groups cannot be provided for each intervention separately, as it was not reported which intervention was being administered at the time the adverse events occurred. Arm 1 refers to the group who received ultrasound-guided injections first and then crossed over to regular injections, and Arm 2 refers to the group who received regular injections and crossed over to ultrasound-guided injections.
Arm/Group | Ultrasound-guided Injections Followed by Regular Injections | Regular Injections Followed by Ultrasound-guided Injections
All-Cause Mortality (participants affected / at risk) | 0/10 | 1/11
Serious Adverse Events (participants affected / at risk) | 0/10 | 0/11
Other Adverse Events (participants affected / at risk) | 0/10 | 1/11
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Ultrasound-guided Injections Followed by Regular Injections (N=10) | Regular Injections Followed by Ultrasound-guided Injections (N=11)
Chest pain (Cardiac disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Small number of subjects analyzed

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No